CLINICAL TRIAL: NCT03594318
Title: Versailles Hospital Cardiac Arrest Registry
Status: Recruiting | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, LEGRIEL stephane, study principal investigator, Versailles Hospital
Other Study IDs: P13/20_ACR
Record Dates: First submitted 2018-07-09; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Out-of-hospital and in-hospital cardiac arrest (CA) requiring intensive care unit management.

Data collection using a standardized form : demographic data and data related to the CA according to the Utstein guidelines.. Circumstances of onset, dates and times of onset and control of abnormal movements (myoclonus and.or seizures).

On-scene clinical findings, pre-hospital and hospital care providers, timing of various treatments and supportive care, results of etiological investigations, cause of CA. Dates and times of EEG monitoring, EEG results. Outcomes including vital status and Cerebral Performance Category scale score at ICU and hospital discharge, day-90 and 1-year after CA and determined based on data in the ICU and/or hospital/neurologist charts and/or general practitionner phone interview.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest requiring Intensive Care Unit management
* Age >= 18 years

Exclusion Criteria:

- Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest requiring Intensive Care Unit Management
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Long term favorable outcome | 1 year
  A favorable outcome is defined by a Cerebral Performance Category scale score (CPC) of 1 or 2. The Cerebral Performance Category scale score will be determined according to hospital charts and/or general practitioner phone interview.
  The CPC score : [5: Death, 4: Persistent vegetative state, 3: Severe disability, 2: Moderate disability, 1 : Low disability]

SECONDARY OUTCOMES:
Short term favorable outcome | 3 months
  A favorable outcome is defined by a Cerebral Performance Category scale score (CPC) of 1 or 2. The Cerebral Performance Category scale score will be determined according to hospital charts and/or general practitioner phone interview.
  The CPC score : [5: Death, 4: Persistent vegetative state, 3: Severe disability, 2: Moderate disability, 1 : Low disability]
Postanoxic Status Epilepticus | 28 days
  Postanoxic Status Epilepticus occurence as defined by EEG abnormalities based on the Salzburg Criteria
Complications of anticoagulant/ antiplatelet therapies | 28 days
  Any bleeding requiring >2 Units Red Blood Cell transfusion
Short term quality of life as assessed by the Short Form (36) Health Survey (SF36) | 3 months
  Description of global SF36 score and each of its eight sections (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health).
Long term quality of life as assessed by the Short Form (36) Health Survey (SF36) | 1 year
  Description of global SF36 score and each of its eight sections (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health).

CONTACTS AND LOCATIONS:
Overall Officials: Legriel Stephane, MD, Study Director — Intensive care unit
Locations (1):
- CH Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No